CLINICAL TRIAL: NCT02728284
Title: Evaluation of Cardiac Function With Cardio-respiratory Synchronized MRI
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-00601
Record Dates: First submitted 2016-03-30; First posted 2016-04-05 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Heart Disease
Keywords: Magnetic Resonance Imaging (MRI)
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Cardiovascular System (Active Comparator): 70 with a history of heart or lung disease
  Interventions: Procedure: cardiovascular MRI (CMR)
- Abnormal Cardiovascular System (Active Comparator): 30 without any history of heart or lung disease
  Interventions: Procedure: Conventional Cardiologic Evaluation

INTERVENTIONS:
Procedure: cardiovascular MRI (CMR) — CMR is used to demonstrate cardiac abnormalities and assess cardiac function in many patients
  Arms: Normal Cardiovascular System
Procedure: Conventional Cardiologic Evaluation — ECG (gating), and respiratory motion effects
  Arms: Abnormal Cardiovascular System

SUMMARY:
The purpose of this investigation is to evaluate newer methods of performing cardiovascular MRI (CMR) that will provide new kinds of information related to the interplay between the cardiac and the respiratory cycles, such as the interaction between the left ventricle and the right ventricle during respiration . The primary statistical objective is to provide preliminary indications of the relative utility of the investigational imaging software in terms of image quality and suitability for routine clinical use. Image quality will be expressed in terms of signal-to-noise ratios (SNR), contrast-to-noise ratios (CNR) and subjective Likert-type qualitative assessments independently provided by each of multiple blinded readers for each image. Suitability for routine use will be assessed in terms of imaging time and a binary indicator of whether, in the opinion of the investigator, adverse procedural complications (not expected) were encountered during a given imaging session.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be selected as they are scheduled for clinical MR examinations.
* Subjects will be selected on the basis of their willingness and ability to participate, on their comprehension of the informed consent document, on their likelihood of completing the study, and on the clinical appropriateness of the investigational technique for a given patient.

Exclusion Criteria:

* electrical implants such as cardiac pacemakers or perfusion pumps
* ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants
* ferromagnetic objects such as jewelry or metal clips in clothing
* pre-existing medical conditions including a likelihood of developing seizures or claustrophobic reactions, and any greater than normal potential for cardiac arrest.

Ages: 7 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-03-29 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Image Quality measured by resolution | 10 Minutes
Image Quality measured by signal to noise | 10 Minutes
Suitability for routine use measured by imaging time and ease of use | 10 Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Leon Axel, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States